CLINICAL TRIAL: NCT04296539
Title: Investigation of the Effect of Regular Exercise on Scapular Muscular Endurance, Scapular Stabilization and Dyskinesia
Brief Title: Compare the Scapular Muscular Endurance, Stabilization and Dyskinesis Parameters of Sedentary Individuals
Status: Completed | Type: Observational
Sponsor: Cyprus International University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sıddıka Fatma Uygur, Professor Doctor PT, Cyprus International University
Other Study IDs: 044-339
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Scapular Dyskinesis; Sedentary Behavior
Keywords: Scapular Dyskinesis; Muscle Strength; Muscle Endurance; Pilates Exercises
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sedentary: Involving little exercise or physical activity
- Exercise: Subjects who were performing regularly pilates exercises for at least six months

SUMMARY:
The aim of this study was to compare the parameters of scapular muscular endurance, scapular stabilization, scapular dyskinesia, upper extremity functional status and postural alignment of adult women aged between 40-65 years old who were performing clinical pilates exercises regularly compared with sedentary adult women in the same age group and to determine whether regular exercise had an effect on these parameters.

DETAILED DESCRIPTION:
The aim of this study was to compare the parameters of scapular muscular endurance, scapular stabilization, scapular dyskinesia, upper extremity functional status and postural alignment of adult women aged between 40-65 years old who were performing clinical pilates exercises regularly compared with sedentary adult women in the same age group and to determine whether regular exercise had an effect on these parameters. A total of 70 individuals were included in the study, including 35 individuals performing regular clinical pilates exercises and 35 individuals with sedentary lifestyles. Clinical pilates group was selected from the individuals who participated in the exercise program under the control of a physiotherapist regularly for 1 hour, 2-3 days a week for at least 6 months. Socio-demographic characteristics, health status and exercise habits of the participants were recorded. For scapular muscle strength assessment, digital hand dynamometer; for scapular muscular endurance assessment, Scapular Muscular Endurance Test (SMET) and Shoulder External Rotation Fatigue Protocol; for the assessment of scapular dyskinesia, Lateral Scapular Slide Test (LSST) and Lennie test; for assessment of upper extremity functional status, Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH); for the assessment of postural alignment, the New York Posture Assessment Test were used.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who perform clinical pilates exercises regularly for at least 6 months and at least 2 days a week (pilates group)
* Individuals who are not actively involved in any sports and do not exercise / physical activity regularly (sedentary group)

Exclusion Criteria:

* Individuals diagnosed with scoliosis or any other orthopedic and neurological problems
* Individuals who have had any diagnosis / treatment or had previous surgery due to shoulder and shoulder circumference problems in the last 6 months
* Individuals with shoulder elevations less than 140 degrees

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 70 Women, 35 Sedentary and 35 Doing Regular Clinical Pilates Exercise
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Scapular Dyskinesia | Twenty minutes
  Scapular Malpositioning, Inferior medial border prominence where the scapula is protracted and is in a anteriorly tilted position.
Scapular muscular endurance | Fifteen minutes
  Repetition and duration of scapular muscles submaximal load

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Ozalp, PhD, Study Chair — Cyprus International University; Baran Yosmaoglu, Professor, Study Chair — Baskent University
Locations (1):
- Cyprus International University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided